CLINICAL TRIAL: NCT05577377
Title: An Unblinded, Uncontrolled, 1-month Interventional Single Group Pilot Study, to Assess the Possibility of Orgasmic Meditation Practice Being Used as a Possible Intervention for PTSD.
Brief Title: OM and Trauma Study
Acronym: OMTP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of OM Foundation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00061665
Record Dates: First submitted 2022-09-29; First posted 2022-10-13 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2022-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Pre and Post Intervention Study with Orgasmic Meditation - a meditation practice
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OM intervention (Experimental)
  Interventions: Behavioral: Orgasmic Meditation

INTERVENTIONS:
Behavioral: Orgasmic Meditation — Orgasmic Meditation (OM) is a structured attention training practice that you do with another person by following a predefined set of detailed instructions. One of the two people participating in the OM must have a clitoris. In this partnered practice, one person strokes the clitoris of another person with the tip of their left index finger for 15 minutes.

SUMMARY:
The primary purpose of this study is to use an unblinded, uncontrolled, 1-month interventional single group pilot study, to assess the possibility of Orgasmic Meditation practice being used as a possible intervention for PTSD. The secondary purpose of this study is to examine if OM is associated with a decrease in the symptoms and self-assessed experiences associated with trauma.

The OM Trauma Protocol (OMTP) is designed to systematize the application of Orgasmic Meditation (OM) for individuals seeking relief from a wide variety of problems and/or help them in their pursuit of eudaimonia. The study protocol will evaluate whether OMing (the act of practicing OM) shows potential for being an effective intervention for people suffering from Post-Traumatic Stress Disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* One or more participants of the pair having a diagnosis of PTSD for > 6 months
* Relationship for > 6 months
* Self or partner of female sex
* Massachusetts residents
* Access and ability to use internet and a video platform called Zoom
* No history of doing the practice of OM

Exclusion Criteria:

* Ongoing or active use of illicit drugs at the time of the study
* Self-identify as pregnant
* Inability to speak English
* Recent hospitalization < 12 months
* Suicidal ideation < 12 months
* Self-harm < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — One of the participant pairs must have a clitoris
Enrollment: 28 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Correlation between OM and PTSD symptoms | 4 weeks
  Change in PCL-5 Score
Number of participants who withdraw from the study | 4 weeks
  Safety will be measured by completion rate
Number of participants who score a 39 or higher using the OM perceived value survey | 4 weeks
  feasibility measured by OM perceived value survey

SECONDARY OUTCOMES:
Correlation between Eudaimonia and OM | 4 weeks
  Changes in Eudaimonia Assessment
Correlation between depression and OM | 4 weeks
  Changes in The Patient Health Questionnaire: Depression Scale (PHQ-9)
Correlation between anxiety and OM | 4 weeks
  Changes in the Generalized Anxiety Disorder 7-Item Scale (GAD-7)
Correlation between psychosocial functioning and OM | 4 weeks
  Changes in The Brief Inventory for Psychosocial Functioning (B-IPF)

OTHER OUTCOMES:
Correlation between OM and tumescence | 4 weeks
  Changes in the Tumescence Assessment. Tumescence is the measure of internal energy available in a person to be used for creativity and purpose

CONTACTS AND LOCATIONS:
Overall Officials: Dan Kriegman, PhD, Principal Investigator — Institute of OM Foundation
Locations (1):
- Institute of OM Foundation, Santa Rosa, California, United States

IPD SHARING:
Plan to Share IPD: No